CLINICAL TRIAL: NCT06705673
Title: Investigation of Gait Profile and Variables of Children and Adolescents with Pediatric Rheumatic Disease Using a Smart Insole System
Brief Title: Gait Profile and Variables in Pediatric Rheumatic Disease Using a Smart Insole System
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Asya Albayrak, MSc, Istanbul Kent University
Other Study IDs: digitsole
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Juvenile Idiopathic Arthritis (JIA); Familial Mediterranean Fever (FMF ); Healthy Controls
Keywords: Juvenile Idıopathic Arthritis; Familial Mediterranean Fever; Gait profile; Smart Insole System; Gait analysis
MeSH Terms: conditions — Arthritis, Juvenile; Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Juvenile Idiopathic Arthritis: Patients diagnosed with JIA who are being followed at the Istanbul Medical Faculty Pediatric Rheumatology Clinic will be included in the study.
- Familial Mediterranean Fever: Patients diagnosed with FMF who are being followed at the Istanbul Medical Faculty Pediatric Rheumatology Clinic will be included in the study.
- Healthy control: For the healthy control group, healthy children and adolescents without any illnesses who volunteer to participate in the study will be included.

SUMMARY:
In pediatric rheumatic diseases, joint swelling, effusion, tenderness, and painful restriction of joint movement, particularly in weight-bearing joints, frequently alter walking function. These changes affect temporal and spatial parameters of gait, as well as kinematic and kinetic characteristics, leading to functional limitations. Comprehensive physical assessments in patients may not always predict changes in gait parameters. Therefore, incorporating objective methods related to gait and balance into physical evaluations is essential for functional insights and clinical decision-making, aiming to prevent adaptive mechanisms that could negatively affect gait function in the long term. In this context, smart insoles have emerged as a new tool for gait analysis, offering an alternative to high-cost, lab-based equipment. The Digitsole Pro® system can measure gait profile and variables in real-life conditions. A review of the literature reveals no studies utilizing smart insole-based gait assessments in pediatric rheumatic patients. The aim of our study is to investigate the gait profile and variables of children and adolescents with pediatric rheumatic disease using the next-generation Digitsole Pro® smart insole system, and to compare the results with those of healthy peers.

ELIGIBILITY:
Inclusion Criteria:

Children and adolescents with pediatric rheumatic disease:

* Aged 6-18 years
* Diagnosed with JIA or FMF at least 6 months ago at the Istanbul Medical Faculty Pediatric Rheumatology Clinic

Healthy children and adolescents:

* Aged 6-18 years
* Willing to participate in the study

Exclusion Criteria:

Exclusion criteria for children and adolescents with pediatric rheumatic disease:

* History of trauma or surgery affecting the musculoskeletal system in the last 6 months
* Presence of a chronic disease other than JIA or FMF
* Acute pain for any reason
* Visual or hearing problems
* Cognitive impairment that prevents understanding of given instructions

Exclusion criteria for healthy children and adolescents:

* History of trauma or surgery affecting the musculoskeletal system in the last 6 months
* Hearing or visual problems
* Acute pain for any reason

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients diagnosed with Juvenile Idiopathic Arthritis (JIA) and Familial Mediterranean Fever (FMF) who are being followed at the Istanbul Medical Faculty Pediatric Rheumatology Clinic will be included in the study. For the healthy control group, healthy children and adolescents without any illnesses who volunteer to participate in the study will be included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-01-06 (Estimated); Study Completion 2025-02-03 (Estimated)

PRIMARY OUTCOMES:
Heel Strike Angle | Baseline
  Monopedal parameters of walking such as heel strike will be assessed with Digitsole Pro.
Heel-Off Angle | Baseline
  Monopedal parameters of walking such as heel-off will be assessed with Digitsole Pro.
Flat Foot | Baseline
  Monopedal parameters of walking such as Flat-Foot (FFI) will be assessed with Digitsole Pro.
Step Length | Baseline
  Monopedal parameters of walking such as step length in meters will be assessed with Digitsole Pro.
Stance Duration | Baseline
  Monopedal parameters of walking such as stance duration time will be assessed with Digitsole Pro.
Percentage of swing time | Baseline
  Monopedal parameters of walking such as percentage of swing time will be assessed with Digitsole Pro.
Cadance | Baseline
  Bipedal parameters of walking such as cadance will be assessed with Digitsole Pro.
Walking speed | Baseline
  Bipedal parameters of walking such as walking speed (km/h) will be assessed with Digitsole Pro.
Double Support Time | Baseline
  Bipedal parameters of walking such as double support time will be assessed with Digitsole Pro.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman, PhD, Principal Investigator — Istanbul University - Cerrahpasa; Asena Yekdaneh, MSc, Principal Investigator — Fenerbahce University; Asya Albayrak, MSc, Principal Investigator — Istanbul University - Cerrahpasa; Fatma Gul Demirkan, Dr, Principal Investigator — Kanuni Sultan Suleyman Eğitim ve Araştırma Hastanesi; Nuray Aktay Ayaz, Prof. Dr., Principal Investigator — Istanbul University

IPD SHARING:
Plan to Share IPD: No